CLINICAL TRIAL: NCT05131815
Title: The BurnAlong Pilot Study: Examining the Feasibility of a Virtual Group-based Physical Activity Intervention for Adolescent and Young Adult Cancer Survivors
Brief Title: The BurnAlong Pilot Study for Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Celina Shirazipour, Assistant Professor, Cancer Research Center for Health Equity, SOCCI, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2020-24-SHIRAZIP-BURN
Record Dates: First submitted 2021-11-02; First posted 2021-11-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Cancer Metastatic; Neoplasms; Breast Cancer; Lung Cancer; Thyroid Cancer; Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Lymphoma; Leukemia; Sarcoma; Skin Cancer; Bone Cancer; Gynecologic Cancer; Pancreas Cancer; Multiple Myeloma; Colorectal Cancer; Gastrointestinal Cancer; Prostate Cancer; Glioblastoma; Brain Cancer; Head and Neck Cancer
Keywords: virtual exercise; adolescent and young adult cancer; BurnAlong App; Well-being; cancer; physical activity
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Lung Neoplasms; Thyroid Neoplasms; Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia; Sarcoma; Skin Neoplasms; Bone Neoplasms; Pancreatic Neoplasms; Multiple Myeloma; Colorectal Neoplasms; Gastrointestinal Neoplasms; Prostatic Neoplasms; Glioblastoma; Brain Neoplasms; Head and Neck Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Group-Based Physical Activity (BurnAlong) and Discussion Board (Experimental): Participants will be asked to complete a 12 week virtual physical activity program delivered by the BurnAlong app, participate in a discussion board, and engage in live physical activity sessions with an exercise physiologist.
  Interventions: Behavioral: Virtual group based physical activity (BurnAlong) and Social Media Discussion Board

INTERVENTIONS:
Behavioral: Virtual group based physical activity (BurnAlong) and Social Media Discussion Board — Participants will engage in two to three virtual physical activity sessions a week through the BurnAlong app for three months with a chosen partner and participate at least twice a week in the research team-mediated social media message board. Additionally, participants will be asked to participate in one live physical activity session per month with an exercise physiologist.

SUMMARY:
The purpose of this prospective, interventional, single-arm pilot study is to evaluate whether virtually delivered group-based physical activity is feasible for adolescent and young adult (AYA) cancer survivors. AYAs who were diagnosed with cancer and have completed cancer treatment will be recruited for this study. This study will enroll 20 participants in total and will last approximately 3 months.

DETAILED DESCRIPTION:
This is a single-arm, prospective, interventional pilot study.

Adolescent and young adult (AYA) survivors of cancer ages 18-39 (n=20) will engage in three months of virtually group physical activity (PA) delivered via BurnAlong, a wellness platform and online app.

Participants will be asked to engage in a BurnAlong workout session with a partner (friend/spouse/child/fellow study participant) a minimum of three times a week for 3 months.

Participants will also meet monthly with an exercise physiologist for a customized exercise session. Participants are allowed to engage in additional PA and non-PA sessions on BurnAlong as desired.

Participants will also be asked to engage in a private social network discussions around key topics of interest for AYA communities with a focus on post-traumatic growth and positive psychology with a minimum of 2 post engagements a week for 3 months.

Participants will complete surveys and physical assessments at baseline and at end of study.

Participants also participate in a 1 hr qualitative exit interview about their well-being, participation experiences, and experience with using the BurnAlong platform.

ELIGIBILITY:
Inclusion Criteria:

* Cancer (all types) diagnosis between the ages of 15-39
* Between the ages of 18-39 during study participation
* At least 3 months post-active treatment completion
* Answers "no" to all questions on the Physical Activity Readiness Questionnaire
* Not currently meeting physical activity guidelines per leisure-time physical activity participation questionnaire
* Access to and ability to use a computer, tablet or phone device with internet access
* Ability to understand and read English
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Hearing loss or vision impairment that would preclude the participant from accessing and using the app (use of hearing aids or visual aids is acceptable) based on self-report
* Currently meeting physical activity guidelines (score of >23 on Godin-Shephard Leisure-Time Physical Activity Questionnaire)
* Currently pregnant, based on self-report
* Patients with active treatment planned within the next 3 months. (Active treatment includes chemotherapy, biologic therapy, radiation therapy, surgery, and any combination.) Long-term hormonal/biologic treatments are acceptable except for AR-targeted therapies for prostate cancer. Participants with known metastatic disease, grade 3 or higher neuropathy, major surgery within 3 months of baseline visit, pregnancy of childbearing potential will be excluded.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of BurnAlong | 12 weeks
  Number of participants that adhere to a 3-month virtually delivered physical activity program via BurnAlong, group discussion boards, and a monthly live physical activity session with an exercise physiologist

SECONDARY OUTCOMES:
Resting Heart Rate | Measured at Baseline and at Week 12
  Evaluate impact of intervention on resting heart rate (bpm) at 3-months (compared to baseline day 0)
Sleep Duration | Measured at Baseline and at Week 12
  Evaluate impact of intervention on sleep duration (number of hours slept each night) at 3-months (compared to baseline day 0)
Sleep Quality | Measured at Baseline and at Week 12
  Evaluate impact of intervention on the percentage of time awake during the night at 3-months (compared to baseline day 0)
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 | Measured at Baseline and at Week 12
  Evaluate short-term effects of virtually delivered exercise, partner support, and group discussion on well-being. PROMIS measures are scored on a T-score metric with a mean of 50 and standard deviation of 10. Scores can be categorized as: within normal limits, mild, moderate and severe.
Post-Traumatic Growth Inventory (PTGI) | Measured at Baseline and at Week 12
  Evaluate short-term effects of virtually delivered exercise, partner support, and group discussion on post-traumatic growth and self-improvement
Health Action Process Approach Inventory (HAPA Inventory) | Measured at Baseline and at Week 12
  Evaluate short-term effects of virtually delivered exercise, partner support, and group discussion on theoretical determinants of physical activity participation as proposed by the Health Action Process Approach (task self-efficacy, outcome expectancies, risk perception, intentions, planning, maintenance self-efficacy, recovery self-efficacy, physical activity behavior) by comparing data at baseline (day 0) and 3 months
Patient-Reported Outcomes Measurement Information System (PROMIS) Social Support | Measured at Baseline and at Week 12
  Evaluate short-term effects of virtually delivered exercise, partner support, and group discussion on social well-being. PROMIS measures of the ability to participate in social roles and activities are scored on a T-score metric with a mean of 50 and standard deviation of 10. Scores can be categorized as: within normal limits, mild, moderate and severe.
Adolescent and Young Adult Psycho-Oncology Screening Tool (AYA-POST) | Measured at Baseline and at Week 12
  Evaluate short-term effects of virtually delivered exercise, partner support, and group discussion on distress and areas of concern such as practical, family, emotional, social, physical, and information
Measure of Experiential Aspects of Participation (MeEAP) | Measured at Baseline and at Week 12
  12 item questionnaire that assesses the 6 experiential aspects of participation (autonomy, belongingness, challenge, engagement, mastery, and meaning) on a 7 point scale (1, strongly disagree, to 7, strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Whiteway, LtCol USAF, MD, Principal Investigator — Walter Reed National Military Medical Center; Celina H Shirazipour, Ph.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: virtual physical activity platform — http://www.BurnAlong.com